CLINICAL TRIAL: NCT00026975
Title: Clinical Outcomes Modeling for Laryngectomy Surgery Patients and Efficacy of Hyperbaric Oxygen Therapy
Brief Title: Efficacy of Hyperbaric Oxygen Therapy in Laryngectomy Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P50AT000428-01P1 (NIH); NCT00052702 (obsolete NCT alias)
Record Dates: First submitted 2001-11-15; First posted 2001-11-16 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Laryngeal Cancer
Keywords: Laryngeal Cancer; Laryngectomy; Tissue Oxygenation; Irradiated Tissue; Hyperbaric Oxygen; Angiogenesis; EF5
MeSH Terms: conditions — Laryngeal Neoplasms | interventions — Hyperbaric Oxygenation

INTERVENTIONS:
Procedure: Hyperbaric Oxygen

SUMMARY:
This study is designed to develop a predictive model for the development of wound complications in patients undergoing laryngectomy surgery for laryngeal/adjoining structure cancers, and to evaluate the clinical efficacy of hyperbaric oxygen for the prevention/management of wound complications in this previously irradiated population. The eligibility profile welcomes the involvement of patients in need of laryngectomies for newly diagnosed cancers and for failed chemoradiation. Patients are afforded the opportunity to be cared for by some of the most distinguished head & neck surgeons and hyperbaric medicine physicians at the University of Pennsylvania in Philadelphia, the oldest teaching medical facility in the country, as well as the Philadelphia Veterans Affairs Medical Center. In addition, participants will be contributing to a body of research uncovering new methods for the assessment of tissue/tumor oxygenation, modeling to promote early wound complication identification, and confirming the role of hyperbaric oxygen therapy in the care and prevention of these problem wounds.

DETAILED DESCRIPTION:
Clinical Outcomes Modeling for Laryngectomy Surgery Patients and Efficacy of Hyperbaric Oxygen Therapy, with Ara Chalian, MD as Project Leader, will develop a predictive model for surgical risk among patients requiring laryngectomy due to cancer, validate the model and assess the efficacy of HB02 therapy for improving outcome. The focus will be to determine the patho-physiological basis for heightened surgical risk among post-radiation head and neck patients and the efficacy of hyperbaric oxygen (HB02) therapy for improving outcome.

This multidisciplinary center will investigate the mechanisms of action, safety, and clinical efficacy of Hyperbaric Oxygen (HB02) Therapy. The group will evaluate if HB02 therapy will benefit patients who must undergo laryngectomy and reconstructive surgery after radiation therapy because, at pharmacological doses, oxygen augments angiogenesis and impedes specific types of intercellular adherence.

The project tests two hypotheses: (1) Predictive models can be developed for sub-groups of head and neck cancer patients who have undergone surgery based on tumor specific site, previous treatment, and co-morbidity and predict which patients will have complications (wound infection and fistula), and (2) HB02 given by a standard protocol can modify tissue hypoxia and vascularity that is present in patients with previous radiation therapy to the neck who have recurrent or secondary cancers requiring laryngectomy. The specific aims are to: (1) develop a detailed database model to predict the risk of developing post-operative complications in complex head and neck aerodigestive tract cancer resections, (2) conduct prospective validation of the predictive model using data on patients treated at the University of Pennsylvania Head and Neck Cancer Center, (3) determine whether hyperbaric oxygen therapy alters post-surgical complication rates and acute and long-term quality of life. The studies include evaluation of clinical parameters, surgical outcome and quality of life measurements, and objective, laboratory-based assessments of the magnitude of hypoxia/vascularization in surgical zones and tumors to provide objective data on surgical risk and clinical responses to HB02 therapy.

The prospective trial allows for planned follow-up and data collection for modeling and tumor oxygenation assessments for patients undergoing laryngectomy. The randomized trial is a treatment trial, comparing standard care before and after laryngectomy to the intervention of pre- & post-operative HBO2 in conjunction with laryngectomy. All patients receive nutritional counseling, speech therapy, and comprehensive peri-surgical care.

ELIGIBILITY:
Inclusion Criteria for Prospective Trial:

* a lesion either suspicious for or diagnosed by biopsy as laryngeal/adjacent pharyngeal cancer requiring a total or partial laryngectomy, or if previously irradiated and ineligible for the randomized trial.
* no history of radiation to the head/neck
* adequate liver and kidney function
* no plans to become pregnant or conceive for the duration of the study

Inclusion Criteria for Randomized Trial:

* have been previously irradiated for a head/neck cancer requiring a total laryngectomy
* demonstrate a lesion either suspicious for or diagnosed by biopsy as laryngeal/adjacent pharyngeal cancer
* have adequate liver and kidney function
* meet physical requirements for hyperbaric oxygen therapy
* agree to randomization of care to receive a laryngectomy and standard follow-up care vs. hyperbaric oxygen therapy preoperatively and postoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2000-09; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Ara A. Chalian, MD, Principal Investigator — Clinical Faculty, Dept. ORLHNS, University of Pennsylvania; Stephen R. Thom, MD PhD, Study Director — Chief of Section, Dept. of Hyperbaric Medicine, University of Pennsylvania
Locations (1):
- University of Pennsylvania Medical Center, Dept.of Otorhinolaryngology, 3400 Spruce Street, 5 Ravdin, Philadelphia, Pennsylvania, United States